CLINICAL TRIAL: NCT06544850
Title: Lateralization Performance and Two-point Discrimination in Patients With Chronic Low Back Pain: A Cross-sectional Study
Brief Title: Lateralization Performance in Chronic Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, Assistant Professor, Inonu University
Other Study IDs: 2024/6004
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low-back Pain
Keywords: pain; rehabilitation; lateralization
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Participants Individuals between 18-65 will be included in the study because pain mechanisms and effects are different between adults and children. Inclusion criteria are having low back pain for 3 months or longer, Mini mental test score>23, Healthy individuals who do not experience chronic low back pain will be evaluated in the control group. Hypertension, congestive heart failure, chronic obstructive pulmonary disease, rheumatological diseases, vertigo, nausea, vomiting, specific diagnosis underlying back pain (e.g. radicular symptoms), significant decrease in vision and hearing, body mass index higher than 30, serious psychiatric condition, inability to communicate, traumatic low back pain, those who have had back surgery, those who refused to participate in the study and did not fill out the consent form will be excluded.
  Interventions: Other: experimental group
- Control Group: Consists of healthy volunteer participants who meet the inclusion criteria. The control group will be selected from those who have never felt back pain that would affect their daily life activities and who have not received treatment.
  Interventions: Other: control group

INTERVENTIONS:
Other: experimental group — Oswestry Low Back Pain Questionnaire will be used to assess functional limitations in daily life activities of patients with low back pain. Recognize mobile application will be used to assess lateralization performance. Evaluation will be made with hand, foot and back modules of this application. Reaction time and accuracy given at the end of the application will be recorded. The most accurate response instruction will be given in the shortest possible time. Visual Analog Scale (VAS) will be used to measure general pain status of patients. Tampa Kinesiophobia Scale will be used to assess fear of movement. Pain catastrophizing level will be assessed with Pain Catastrophizing Scale. Two-point discrimination device will be used to assess two-point discrimination. Central Sensitization Inventory will be used for central sensitization findings.
  Groups: Experimental Group
Other: control group — Healthy volunteer participants who meet the inclusion criteria will be evaluated with the tests applied to the experimental group
  Groups: Control Group

SUMMARY:
The aim of our study was to examine the relationship between lateralization performance, two-point discrimination, kinesiophobia and pain catastrophizing in patients with chronic low back pain.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria and agree to participate in the study will be selected from the relevant population by the improbable random sampling method. Demographic data, age, gender, height, weight), education status, and dominant hand and foot information will be obtained from the volunteer participants participating in the study before starting the study. Oswestry Low Back Pain Questionnaire will be used to evaluate functional limitations in daily life activities of patients experiencing low back pain. This questionnaire has 6 sections with 0-5 points for each question. It consists of 10 sections including pain intensity, personal precautions, lifting objects, walking, sitting, standing, sleeping, sexual life, social life, and travel. 0-4 points are considered as no disability, 5-14 points as mild, 15-24 points as moderate, 25-34 points as severe, and 35-50 points as complete disability. The minimum score received from the scale is 0 and the maximum score is 50. A score of 50 indicates the highest level of functional disability . Recognize mobile application will be used to evaluate lateralization performance. This application will be evaluated with the hand, foot and back modules. The photographs will be shown on a screen. If the patient thinks the photo belongs to the right side, the patient will press the right button and if the patient thinks the photo belongs to the left side, the patient will press the left button. The reaction time and accuracy given at the end of the application will be recorded. The most accurate response instruction will be given in the shortest possible time. The Visual Analog Scale (VAS) will be used to measure the general pain status of the patients. In addition, the duration of the pain, the localization of the pain (right, left) and the Tampa Kinesiophobia Scale will be used to evaluate the fear of movement. This scale consists of 17 items. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement. Each item is scored on a 4-point Likert scale (1-4). The answers and their numerical values are as follows: (1) I strongly disagree, (2) I disagree, (3) I agree and (4) I strongly agree. The scores of items 4, 8, 12 and 16 should be reversed when calculating the total score. The total score obtained by adding different items can vary between 17-68. The level of pain catastrophizing will be assessed with the Pain Catastrophizing Scale. This scale is a 5-point Likert-type scale consisting of 13 questions and evaluates the feelings and thoughts of the person when experiencing pain. A two-point discrimination device will be used to assess two-point discrimination. The Central Sensitization Inventory will be used for central sensitization findings. Part A, consisting of 25 items scored from 0 to 4, will be used. A higher score indicates the presence of more symptoms related to central sensitization. A cut-off value equal to or above 40 indicates the presence of central sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain for 3 months or longer
* Mini mental test score>23
* Healthy individuals in the control group who do not have chronic low back pain

Exclusion Criteria:

* Hypertension
* chronic obstructive pulmonary disease
* specific diagnosis underlying back pain (e.g. radicular symptoms)
* inability to communicate
* those who refused to participate in the study and did not fill out the consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy individuals and participants with chronic low back pain
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Lateralization Performance | 4 months
  The Recognize mobile application will be used to evaluate lateralization performance. The evaluation will be made with the hand, foot and back modules of this application. The photos will be shown on a screen. If the photo is from the right side, the person will press the right button and if it is from the left side, the person will press the left button. The reaction time and accuracy given at the end of the application will be recorded. The most accurate response instruction will be given in the shortest possible time

SECONDARY OUTCOMES:
Oswestry Disability Index | 4 months
  Oswestry Low Back Pain Questionnaire will be used to evaluate functional limitations in daily life activities of patients with low back pain. This questionnaire has 6 sections with scores ranging from 0 to 5 for each question. It consists of 10 sections including pain intensity, personal precautions, lifting objects, walking, sitting, standing, sleeping, sexual life, social life, and travel. 0-4 points are considered as no disability, 5-14 points as mild, 15-24 points as moderate, 25-34 points as severe, and 35-50 points as complete disability. The minimum score received from the scale is 0 and the maximum score is 50. A score of 50 indicates the highest level of functional disability
Visual Analogue Scale | 4 months
  Visual Analog Scale (VAS) will be used to measure the general pain status of the patients. In addition, the duration of the pain, the localization of the pain (right, left)
Tampa Scale of Kinesiophobia | 4 months
  The Tampa Kinesiophobia Scale will be used to assess fear of movement. This scale consists of 17 items. A high score indicates a high level of fear of movement, while a low score indicates a negligible level of fear of movement. Each item is scored on a 4-point Likert scale (1-4). The answers and their numerical values are as follows: (1) strongly disagree, (2) disagree, (3) agree, and (4) strongly agree. The scores of items 4, 8, 12, and 16 should be reversed when calculating the total score. The total score obtained by adding the different items can vary between 17-68.
Central Sensitization inventory | 4 months
  For central sensitization findings, the Central Sensitization Inventory will be used. Part A, consisting of 25 items scored from 0 to 4, will be used. A higher score indicates the presence of more symptoms associated with central sensitization. A cut-off value equal to or above 40 indicates the presence of central sensitization
Pain Catastrophizing Scale | 4 months
  The level of pain catastrophizing will be assessed with the Pain Catastrophizing Scale. This scale is a 5-point Likert-type scale consisting of 13 questions and evaluates the feelings and thoughts of the person when experiencing pain
Two Point Discrimination | 4 months
  A two-point discrimination device will be used to evaluate two-point discrimination

CONTACTS AND LOCATIONS:
Overall Officials: YÜKSEL, Principal Investigator — Assistant researcher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsay A, Allen TJ, Proske U, Giummarra MJ. Sensing the body in chronic pain: a review of psychophysical studies implicating altered body representation. Neurosci Biobehav Rev. 2015 May;52:221-32. doi: 10.1016/j.neubiorev.2015.03.004. Epub 2015 Mar 14. PMID 25783221